CLINICAL TRIAL: NCT02522637
Title: What is the Best Frequency of Exercise Training in Severe COPD?
Brief Title: Exercise Training in Severe COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Collaborators: Villa Pineta Hospital (Other)
Responsible Party: Principal Investigator, Mara Paneroni, Physical therapist, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fondazione Salvatore Maugeri
Record Dates: First submitted 2015-07-06; First posted 2015-08-13 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COPD
Keywords: exercise; training; endurance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training F1 (Active Comparator): Patients will be treated with a specific rehabilitation in-hospital program consisting of one daily sessions of 30 minutes of exercise (Frequency 1 : Program F1 )
  Interventions: Other: Exercise training
- Exercise training F2 (Experimental): Patients will be treated with a specific rehabilitation in-hospital program consisting of two daily sessions of 30 minutes of exercise (Frequency 2 : Program F2 )
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — The workout will start with a workload of 50% of the theoretical maximum Watts indirectly assessed by the 6-Minutes Walking Test (6MWT) with equation of Luxton et al. Each training session will begin with three minutes of warm-up and cool-down with a low load.
  At the end of each session, the physiotherapist will administer the Borg Scale (i.e. for dyspnea and muscle fatigue) and detect the oxygen saturation. The sessions will be conducted at constant load for 25 minutes and increase following the Maltais protocol (the workload increase in the next session will be 10 W, if dyspnea and muscle fatigue, evaluated at the Borg Scale, were each < 5 ).
  The patients will perform a supervised 20-min light warm-up gym exercise before the endurance training session. The training will be carried out with the oxygen level necessary to maintain the saturation level ≥ 91%.

SUMMARY:
International guidelines for pulmonary rehabilitation describe pathways dedicated to moderate COPD patients looking at the work setting, programs and frequency of training sessions in an outpatient program of rehabilitation. However, a new population of respiratory patients is growing: these are more serious and older patients, with several comorbidities and recurrent hospitalizations. In this population no guidelines are available to describe the optimum prescription in terms of frequency, intensity, type and timing (FITT) of rehabilitation. In this kind of patients, only few studies are available on the overtraining risk. The aims of the current study are:

1. To detect and compare the response in terms of endurance of two endurance training programs with different time-frequencies (1 session / day versus 2 sessions / day) during 30 days of in-hospital admission to a pulmonary rehabilitation center
2. To compare the effectiveness in terms of effort tolerance, dyspnea, peripheral and respiratory muscle strength, quality of life and psychological and functional impact of the disease.

DETAILED DESCRIPTION:
Rehabilitation in-hospital program

The rehabilitation program (RP) will start the day after the in-hospital admission and will be continuously supervised by a physiotherapist. The patients will use the drugs and the oxygen therapy prescribed. RP will include a training session on cycloergometer at constant load once a day (Group F1) or twice-a day (Group F2) interrupted by at least three hours of rest. The workout will start with a workload of 50% of the theoretical maximum Watts indirectly assessed by the 6-Minutes Walking Test (6MWT) with equation of Luxton et al.

Measures

At baseline (T0) we will gather in both groups the following evaluations:

1. Anthropometric parameters (age, BMI)
2. Scale of comorbidity CIRS

At the baseline (T0) and end of the program (T1) we will collect, in all patients, the following evaluations:

1. 6-minute walking test walk (6MWT) will be performed according to international guidelines. In patients using oxygen during walking, the oxygen flow will be adjusted to increase the oxygen saturation over 96%.The 6MWT at T1 will be performed with the same amount of oxygen used in the initial test (T0).
2. Endurance cycloergometer test will be performed at 80% of Watts max predicted by the 6MWT. At the beginning, the test will be performed at charge "zero watts" for 2 minutes, then the workload will be increased to 80% of the theoretical max Watts until muscle exhaustion (Borg score > 8), presence of high dyspnea (Borg score > 8) or the achievement of 90% of theoretical maximal heart rate. The final endurance test will be repeated at the same load (speed 50-60 rpm). The time spent for performing the exercise will be registered. In a subset of patients (belonging to the Institute of Lumezzane) the endurance cycloergometer test on the quadriceps muscle will be executed by the Near Infrared Spectroscopy (NIRS ).
3. Scale of the MRC dyspnea
4. Arterial blood gas analysis
5. Respiratory muscle strength (Maximal lnspiratory Pressure [MIP] and Maximal Espiratory Pressure [MEP])
6. Biceps and quadriceps muscle strength evaluated with dynamometer manual
7. CAT scale

Only at the end of the program (T1) we will collect:

1. patient satisfaction by a Likert scale taking into consideration the quantity, quality, and impact of rehabilitation on hospitalization
2. The time consuming for the two programs
3. The side effect
4. The drop out (waste, flare)

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 80 years
* Diagnosis of moderate to severe COPD ( GOLD III and IV ) with clinical stability ( pH> 7.38 and no need to change prescription of respiratory drugs in the last 10 days).

Exclusion Criteria:

* Patients with respiratory failure in absence of COPD
* Patients who had attended a pulmonary rehabilitation program in the last 6 months
* Patients with a recent myocardial infarction (in the last 3 months)
* Patients with congestive heart failure
* Patients with severe orthopedic diseases
* Patients with psychiatric illness and severe cognitive impairment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Endurance cycloergometer test: difference between F1 and F2 programs (time needing for the test execution) | 30 days
  Evaluation of the time needing for the test execution

CONTACTS AND LOCATIONS:
Overall Officials: Mara Paneroni, PT, Principal Investigator — Fondazione Salvatore Maugeri
Locations (1):
- Fondazione Salvatore Maugeri, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Publication

REFERENCES:
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Luxton N, Alison JA, Wu J, Mackey MG. Relationship between field walking tests and incremental cycle ergometry in COPD. Respirology. 2008 Nov;13(6):856-62. doi: 10.1111/j.1440-1843.2008.01355.x. PMID 18811884
- [Background] Brooks D, Solway S, Gibbons WJ. ATS statement on six-minute walk test. Am J Respir Crit Care Med. 2003 May 1;167(9):1287. doi: 10.1164/ajrccm.167.9.950. No abstract available. PMID 12714344
- [Background] Hook JL, Arcasoy SM, Zemmel D, Bartels MN, Kawut SM, Lederer DJ. Titrated oxygen requirement and prognostication in idiopathic pulmonary fibrosis. Eur Respir J. 2012 Feb;39(2):359-65. doi: 10.1183/09031936.00108111. Epub 2011 Sep 1. PMID 21885386
- [Result] Paneroni M, Vogiatzis I, Belli S, Savio G, Visca D, Zampogna E, Aliani M, Carolis V, Maniscalco M, Simonelli C, Vitacca M. Is Two Better Than One? The Impact of Doubling Training Volume in Severe COPD: A Randomized Controlled Study. J Clin Med. 2019 Jul 18;8(7):1052. doi: 10.3390/jcm8071052. PMID 31323895